CLINICAL TRIAL: NCT02824302
Title: A Prospective Observational Study to Evaluate Efficacy of Simple Questions to Predict Labor Pain and Epidural Analgesia Use in Parturients
Brief Title: 3 Simple Questions to Predict Labor Pain and Epidural Analgesia Use in Parturients
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 107817
Record Dates: First submitted 2016-05-13; First posted 2016-07-06 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Survey — Patients coming for induction of labor will be handed a survey regarding their expectation of their coming labor pain. And then will be followed up after 24 hours of their delivery.

SUMMARY:
Labor pain is complex to understand and challenging to define because of the interaction of multiple maternal and fetal factors. Poorly controlled acute post-procedural pain may result in harmful physiological and psychological consequences for both mother and baby. It is therefore important to understand the prelabor factors that may affect the labour pain to facilitate the intrapartum pain management. The goal of this prospective observational study is to verify if expectations regarding pain experience translate to actual pain outcomes for women who are undergoing induction of labor.

DETAILED DESCRIPTION:
A prospective observational cohort study. 100 parturients having induction of labor that match inclusion criteria will be asked to participate. After written informed consent, vital signs and patient demographics will be obtained and recorded. A 3 question survey will be given. Patients will be asked to rate, using a 0-10 cm visual analog scale (VAS), their anxiety level ("On a scale of 0-10 cm, with 0 being not anxious at all through 10 being extremely anxious, how anxious are you about your upcoming labor and delivery?"), their anticipated pain ("On a scale of 0-10, with 0 being no pain at all and 10 being pain as bad as you can imagine, how much pain do you anticipate experiencing during your upcoming labor and delivery?"), and using a categorical scale, to rate their anticipated epidural analgesic need ("On a scale of 0-5, with 0 being none at all, 1 being much less than average, 2 being less than average, 3 being average, 4 being more than average, and 5 being much more than average, how much epidural pain medication do you anticipate needing during your upcoming labor and delivery?"). Then 24 hours after delivery, patient VAS scores will be recorded, number of boluses, total number of hours of labor, patient comfort level and satisfaction

ELIGIBILITY:
Inclusion criteria:

1. The patient is 18 years or older
2. ASA class II or III according to the 2014 American Society of Anesthesiologists' physical status classification
3. The patient is having induction of labor
4. The patient is having a singleton pregnancy
5. the fetus's gestational age is more than 37 weeks
6. the patient is considering having epidural analgesia.

Exclusion criteria:

1. The patient has refused to participate
2. There is a language barrier between the patient and the investigator
3. The patient received narcotics within the last two hours
4. the patient has chronic pain issues
5. There is significant concern about maternal or fetal welfare
6. The patient has a history of opioid tolerance
7. The patient has major psychiatric problem,
8. There is contraindication to epidural labor analgesia
9. Patient has allergy to local anesthetics.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy full term pregnant patients with singleton pregnancy
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | this outcome will measure the pain scores during labour from the start of epidural insertion until its discontinued.
  this outcome will be measured at day 1 of delivery

SECONDARY OUTCOMES:
Time from onset of labor to epidural analgesia | minutes > 30 minutes
Cervical dilatation at the time of request(cm) | hours (>1 hour)
Pain score at the time of request of labor analgesia | VAS (1-10)
Duration labor | hours (> 1 hour)
Number of epidural boluses | hours (> 1 hour)
Patient comfort during labor (1-5) | hours (>1 hour)
Pain VAS during Epidural insertion (0-10) | hours (> 1 hour)
Patient satisfaction with epidural analgesia | hours ( >1 hour)
Mode of delivery | hours (>1 hour)

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Science Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Pan PH, Tonidandel AM, Aschenbrenner CA, Houle TT, Harris LC, Eisenach JC. Predicting acute pain after cesarean delivery using three simple questions. Anesthesiology. 2013 May;118(5):1170-9. doi: 10.1097/ALN.0b013e31828e156f. PMID 23485992
- [Result] Carvalho B, Zheng M, Harter S, Sultan P. A Prospective Cohort Study Evaluating the Ability of Anticipated Pain, Perceived Analgesic Needs, and Psychological Traits to Predict Pain and Analgesic Usage following Cesarean Delivery. Anesthesiol Res Pract. 2016;2016:7948412. doi: 10.1155/2016/7948412. Epub 2016 Apr 7. PMID 27143966
- [Result] Carvalho B, Zheng M, Aiono-Le Tagaloa L. A prospective observational study evaluating the ability of prelabor psychological tests to predict labor pain, epidural analgesic consumption, and maternal satisfaction. Anesth Analg. 2014 Sep;119(3):632-640. doi: 10.1213/ANE.0000000000000357. PMID 25029661